CLINICAL TRIAL: NCT04158570
Title: Role of Nephrolithometric Scoring Systems in Prediction of Percutaneous Nephrolithotomy Outcomes in Adult
Brief Title: Role of Nephrolithometric Scoring Systems in Prediction of PCNL Outcomes in Adult
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ehab Abdelwahab Desoky Abdelmoniem, Dr Ehab EL Desoky urology specialist, Assiut University
Other Study IDs: renal stones classification
Record Dates: First submitted 2019-11-01; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Upper Urinary Tract Stones
MeSH Terms: conditions — Urinary Calculi | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous Nephrolithotomy — Application of different stone scoring systems :
  * Guy's scoring system (GSS).
  * Seoul renal stone complexity scoring system (S-ReSC).
  * S.T.O.N.E. nephrolithometry scoring system.
  * CROES Nomogram. These scoring systems will be applied on each patient and correlate the predictive values with the real results to know which one of the above scoring systems better predict the outcomes.

SUMMARY:
Prospective study is to compare between different nephrolithometric scoring systems in prediction of PCNL outcomes in terms of efficacy , success rate and safety in Adult patients with UUT stones unilateral or bilateral, single or multiple, Pelvic or calyceal, primary or recurrent, both gender attending Assuit Urology & Nephrology University Hospital.

DETAILED DESCRIPTION:
The incidence of urolithiasis is approximately 5% to 10% in the general population, In an active urologic department, 30% of the surgical working load is known to be related to treatment of renal and ureteral stones (1, 2). Since the original description of stone removal through a percutaneous nephrostomy tract by Fernstrom and Johansson in 1976, percutaneous stone removal has evolved into a highly developed procedure practiced by many urologists (3). Several new techniques and technologies recently have emerged that simplified the procedure, allowed to take on more challenging cases and made it safer and less painful for patients (4).

Nephrolithometric scoring systems have been introduced to overcome limitations for systematic and quantitative assessment of the outcomes of PCNL. Moreover, preoperative patient counselling necessitates the development of an integrated scoring system to assess PCNL complexity for optimal decision-making Nephrolithometric scoring systems include the Guy's Stone Score (5), S.T.O.N. E. (Stone Size, Tract length, Obstruction/hydronephrosis, Number of involved calyces, Essence/Hounsfield units) nephrolithometry scoring system (6), The Clinical Research Office of the Endourology Society (CROES) nomogram (7), and the Seoul National University Renal Stone Complexity (S-ReSC) score (8,9). All these nephrolithometry scoring systems (NLSS) aim for preoperative prediction of stone-free status (SFS) and complications through assessment of the complexity of different cases undergoing PCNL. NLSS do not only consider the imaging criteria of stones and renal anatomy, but also relevant patient characteristics such as body mass index, previous renal surgery, and surgeon experience. The Guy's Stone Score, S.T.O.N.E. nephrolithometry score and CROES nomogram consist of 11 variables, including four shared parameters (stone size, location, number, and staghorn status). Other variables which are considered by these three NLSS are stone density, renal anatomy, tract length, obstruction of renal pelvis, case load/year, prior treatment history, and the presence of spina bifida or spinal injury.

The Guy's Stone score categorises PCNL cases into four grades, increasing in complexity from Grade 1 to Grade 4, depending on patients' past medical history and non-contrast CT (NCCT) (5).

The S.T.O.N.E. nephrolithometry scoring system assesses PCNL complexity by nine different possible scores, ranging from 5 to 13, according to five NCCT-calculated parameters including stone size, tract length, obstruction/ hydronephrosis, number of involved calyces, Essence/ Hounsfield units (6).

the CROES nephrolithometric nomogram predicts treatment success using plain X-ray of the kidneys, ureters and bladder considering the stone burden, count, and location, in addition to case volume and prior stone treatment (7).

The total score to predict the chance of treatment success is the sum of individual scores derived from each predicting variable; the higher the score, the higher the chance of treatment success, while a patient with a low score has a low chance of achieving a SFS (7). On the other hand, the S-ReSC score is calculated by counting the number of sites involved in the renal pelvis and calyces, regardless of stone parameters or renal anatomy. This system assigns a score from 1 to 9 depending mainly on the number of sites involved; the renal pelvis (1), superior and inferior major calyces (2-3), anterior and posterior minor calyces of the superior (4-5), middle (6-7), and inferior calyces (8-9).

ELIGIBILITY:
Inclusion criteria:

* Adult Patients with renal stones scheduled for PCNL.

Exclusion criteria:

* uncorrected coaguloapathy
* skeletal deformities affect lithotomy position
* Pregnancy.
* Patients <16yr.

Ages: 17 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: no description
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-11-25 (Estimated); Study Completion 2021-11-25 (Estimated)

PRIMARY OUTCOMES:
stone clearance | 1 or 2 day postoperatively
  postoperative stone and CT-KUB will be done to evaluate the presence of stones .

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Hospital, Asyut, Egypt